CLINICAL TRIAL: NCT02119416
Title: Sex and Pubertal Stage Differences in Cardiovascular Responses to Caffeine in Children
Brief Title: Gender Difference in Response to Caffeine in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jennifer Temple, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R01DA030386 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Cardiovascular influences; caffeine; healthy children
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1mg/kg Caffeine (Experimental): Order of Caffeine Administration for Visits 1-6: 1mg, 2mg, 0mg, 1mg, 2mg, 0mg
  Interventions: Drug: Low Caffeine Administration first (1mg/kg body weight)
- 2mg/kg caffeine (Experimental): Order of Caffeine Administration for Visits 1-6: 2mg, 0mg, 1mg, 2mg, 0mg, 1mg
  Interventions: Drug: High Caffeine Administration first (2mg/kg body weight)
- Placebo (Experimental): Order of Administration for Visits 1-6: 0mg, 1mg, 2mg, 0mg, 1mg, 2mg
  Interventions: Drug: Placebo Administration first

INTERVENTIONS:
Drug: Placebo Administration first — All participants received each dose on two days and the order of administration was counterbalanced.
  Order of Administration for Visits 1-6: 0mg, 1mg, 2mg, 0mg, 1mg, 2mg
  Arms: Placebo
Drug: Low Caffeine Administration first (1mg/kg body weight) — On two of the 6 visits, participants received a placebo (flattened sprite) added to their beverage.
  Order of Caffeine Administration for Visits 1-6: 1mg, 2mg, 0mg, 1mg, 2mg, 0mg
  Arms: 1mg/kg Caffeine
Drug: High Caffeine Administration first (2mg/kg body weight) — On two of the 6 visits, participants received a placebo (flattened sprite) added to their beverage.
  Order of Caffeine Administration for Visits 1-6: 2mg, 0mg, 1mg, 2mg, 0mg, 1mg
  Arms: 2mg/kg caffeine

SUMMARY:
Caffeine use is on the rise in America, and one of the most popular sources is soda. Among youth ages 8-16, caffeine consumption has increased by over 70% in the past 30 years. Few studies have examined the role of hormones in caffeine consumption within this age group.

The purpose of the current experiment was to determine the effect of caffeine on children 8 and 9 compared to those 15 and 16 years of age. The investigators were looking at the effect of puberty on the consumption of caffeine as well as the effect that the caffeine has on the body (for example: heart rate, blood pressure) and cognitive function.

DETAILED DESCRIPTION:
Our previous studies have demonstrated sex differences in both the reinforcing properties of (Temple JL, Briatico LN, Clark EN, Dewey AM, 2009) and physiological responses to (Temple JL, Dewey AM, Briatico LN, 2010) caffeine. This is consistent with the literature on other types of drugs showing that men and women often differ in both drug self administration (Lynch WJ,2008 ) and drug sensitivity (Temple, JL, et al, 2008). These differences have been attributed, at least in part, to differences in gonadal hormones (Lynch WJ, 2008) ,Dreher JC et al, 2007). Our laboratory conducted a study investigating subjective effects of caffeine in post-pubertal adolescents and found that boys reported greater drug effects and liking of drug effects than did females (Temple JL, Dewey AM, Briatico LN, 2010, Temple JL, Ziegler AM,2011). In addition, the differences in feeling of the drug effects were related to salivary estradiol levels in females, but not in males, suggesting that steroid hormones can mediate the subjective effects of caffeine. When taken together, these data suggest that there are gender differences in acute and chronic effects of caffeine and that these differences may be mediated by differences in circulating steroid hormones. Previous studies have shown that subjective responses to caffeine vary across the menstrual cycle (Terner JM, de Wit H, 2006), with the greatest subjective effects occurring during the follicular phase, when estradiol levels begin to rise and peak just prior to the ovulatory LH surge. To date, no well-controlled studies have been conducted in humans examining the relationship between steroid hormones and caffeine effects on cognition, which the investigators will address in this study.

ELIGIBILITY:
Inclusion Criteria:

* males and females from 8-9 yoa or 15-17 yoa (post pubertal)
* those 8-9 much have Tanner Staging below 3
* those 15-17 much have Tanner Staging above 3.
* willing to come into the lab 6 times for 1.5-2 hours each
* those willing to abstain from consuming caffeine for 24 hours before each appointment
* those willing to withdraw from consuming anything other than water for 2 hours before each appointment.
* 15-17 year old females much have begun menarche

Exclusion Criteria:

* those on ADHD medication or other's impacting caffeine metabolism
* those reporting being on birth control or other hormones
* those that are pregnant or breastfeeding
* those outside the given age range or pubertal classification
* those reporting having an adverse effect of caffeine in the past

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Temple, PhD, Principal Investigator — SUNY Buffalo; Amanda M Ziegler, MPH, Study Director — SUNY Buffalo; Adam M Graczyk, MS, Study Director — SUNY Buffalo
Locations (1):
- State University at New York at Buffalo, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1mg/kg Caffeine: Order of Caffeine Administration for Visits 1-6: 1mg/kg then 2mg/kg then 0mg/kg
- 2mg/kg Caffeine: Order of Caffeine Administration for Visits 1-6: 2mg/kg then 0mg/kg then 1mg/kg
- Placebo: Order of Administration for Visits 1-6: 0mg/kg then 1mg/kg then 2mg/kg
Period: Overall Study
Arm/Group | 1mg/kg Caffeine | 2mg/kg Caffeine | Placebo
Started | 32 | 36 | 33
Completed | 30 | 35 | 31
Not Completed | 2 | 1 | 2
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — wrong pubertal stage | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: all participants had all treatments across all studies on this project
Groups:
- Total: Total of all reporting groups
Arm/Group | 1mg/kg Caffeine | 2mg/kg Caffeine | Placebo | Total
Number analyzed (Participants) | 30 | 35 | 31 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 35 | 31 | 96
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (1.1) | 12.2 (1.1) | 12.2 (1.1) | 12.2 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 14 | 44
  Male | 17 | 18 | 17 | 52
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 31 | 96

OUTCOME MEASURES:

1. Primary Outcome: Peak Heart Rate After 2 mg/kg of Caffeine
Description: Heart rate measurements were taken every 10 minutes, following 1 minute of rest with an automated Welch Allen Blood Pressure Cuff. We have reported the data as the peak heart rate after 2 mg/kg.
Time Frame: Heart rate was collected every 10 minutes for 60 minutes after the dose of caffeine.
Measure: Mean (Standard Error); unit: beats per minute
Groups:
- 1mg/kg Caffeine Then 2 mg/kg Then 0 mg/kg: Order of Caffeine Administration for Visits 1-6: 1mg/kg then 2mg/kg then 0mg/kg
- 2mg/kg Caffeine Then 0 mg/kg Then 1 mg/kg: Order of Caffeine Administration for Visits 1-6: 2mg/kg then 0mg/kg then 1mg/kg
- 0 mg/kg Then 1 mg/kg Then 2 mg/kg: Order of Administration for Visits 1-6: 0mg/kg then 1mg/kg then 2mg/kg
Arm/Group | 1mg/kg Caffeine Then 2 mg/kg Then 0 mg/kg | 2mg/kg Caffeine Then 0 mg/kg Then 1 mg/kg | 0 mg/kg Then 1 mg/kg Then 2 mg/kg
Number analyzed (Participants) | 30 | 35 | 31
beats per minute | 73.6 (2.32) | 73.2 (1.6) | 79.6 (2.64)
Statistical Analysis 1: Comparison: 1mg/kg Caffeine Then 2 mg/kg Then 0 mg/kg vs 2mg/kg Caffeine Then 0 mg/kg Then 1 mg/kg vs 0 mg/kg Then 1 mg/kg Then 2 mg/kg; Test type: Other — Maximum heart rate after 2 mg/kg of caffeine compared to baseline was assessed using a mixed effects regression model. Sex and pubertal stage were included in the model as time invariant predictors; p < 0.05, mixed effects regression — The p-value was not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: 1mg/kg Caffeine Then 2 mg/kg Then 0 mg/kg vs 2mg/kg Caffeine Then 0 mg/kg Then 1 mg/kg vs 0 mg/kg Then 1 mg/kg Then 2 mg/kg; We used repeated measures ANOVAS and conducted planned comparisons between groups as post-hoc tests; Test type: Other — We compared means of our dependent variables after administration of different doses of caffeine; p < 0.05, ANCOVA — The p-value was set prior to the analysis and all comparisons were planned

2. Primary Outcome: Peak Systolic Blood Pressure
Description: Blood pressure measurements were taken every 10 minutes, following 1 minute of rest with an automated Welch Allen Blood Pressure Cuff. We have reported the peak heart rate after the 2 mg/kg dose of caffeine.
Time Frame: Blood pressure was assessed every 10 minutes for 60 minutes after caffeine was administered.
Population: Participants were randomized to a particular order, but this was a crossover design.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- 1mg/kg Caffeine Then 2 mg/kg Than 0 mg/kg: Order of Caffeine Administration for Visits 1-6: 1mg/kg then 2mg/kg then 0mg/kg
- 2mg/kg Caffeine Than 0 mg/kg Than 1 mg/kg: Order of Caffeine Administration for Visits 1-6: 2mg/kg then 0mg/kg then 1mg/kg
- 0 mg/kg Than 1 mg/kg Than 2 mg/kg: Order of Administration for Visits 1-6: 0mg, 1mg, 2mg, 0mg, 1mg, 2mg
  Placebo Administration first: All participants received each dose on two days and the order of administration was counterbalanced.
  Order of Administration for Visits 1-6: 0mg, 1mg, 2mg, 0mg, 1mg, 2mg
Arm/Group | 1mg/kg Caffeine Then 2 mg/kg Than 0 mg/kg | 2mg/kg Caffeine Than 0 mg/kg Than 1 mg/kg | 0 mg/kg Than 1 mg/kg Than 2 mg/kg
Number analyzed (Participants) | 30 | 35 | 31
mmHg | 107.6 (1.82) | 112.3 (1.69) | 109.6 (2.09)
Statistical Analysis 1: Comparison: 1mg/kg Caffeine Then 2 mg/kg Than 0 mg/kg vs 2mg/kg Caffeine Than 0 mg/kg Than 1 mg/kg vs 0 mg/kg Than 1 mg/kg Than 2 mg/kg; order was included in the analysis. We examined caffeine dose; Test type: Other — mixed effects regression models were used with sex and pubertal stage as time invariant predictors; p < 0.05, mixed effects regression
Statistical Analysis 2: Comparison: 1mg/kg Caffeine Then 2 mg/kg Than 0 mg/kg vs 2mg/kg Caffeine Than 0 mg/kg Than 1 mg/kg vs 0 mg/kg Than 1 mg/kg Than 2 mg/kg; Test type: Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: We collected adverse events over the five year period covered by this funding proposal.
Arm/Group | 1mg/kg Caffeine | 2mg/kg Caffeine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/96 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96 | 0/96
Other Adverse Events (participants affected / at risk) | 0/96 | 0/96 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No